CLINICAL TRIAL: NCT04182789
Title: A Prospective Single Arm Exploratory Clinical Research on the Efficacy and Safety of KN035 in Patients With Advanced Multiple Primary Tumors
Brief Title: KN035 in Patients With Advanced Multiple Primary Tumors
Acronym: CPOG035-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Haiyan Yang, ONCOLOGY DEPT., RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHY
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Multiple Primary Neoplasm
MeSH Terms: conditions — Neoplasms, Multiple Primary | interventions — envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN035 (Experimental): KN035150mg，once a week, subcutaneously. Every 28 days is a treatment cycle.KN035 can be used for up to 2 years.
  Interventions: Drug: KN035

INTERVENTIONS:
Drug: KN035 — KN035150mg，once a week, subcutaneously. Every 28 days is a treatment cycle.KN035 can be used for up to 2 years.

SUMMARY:
This study is a prospective, single arm, single center exploratory clinical research, to evaluate KN035 late treatment in patients with Multiple Primary tumors (MPC, Multiple Primary working) clinical benefit.In the study, all subjects meeting the criteria for inclusion will be enrolled in the KN035 treatment group, and patients cannot receive any other anti-tumor treatment during the study period.The primary endpoint of the study was defined as patients who could be assessed by imaging, and the optimal Objective Response Rate (ORR) based on RECIST 1.1 standard, while the secondary endpoint was safety (nci-ctcae 4.0), DCR (Disease Control Rate), DoR (Duration of Response), progression-free survival (PFS),1) Overall Survival and Overall Survival;The end point of the exploratory study was the correlation between different molecular types and the efficacy of immunotherapy.

DETAILED DESCRIPTION:
Patients diagnosed with advanced MPC in the study should be enrolled as:

Histopathological diagnosis of multiple primary tumors, and is currently suffering from advanced colorectal cancer;Except for bowel cancer, no anti-tumor treatment is needed for other tumors during screening.

The maximum time interval between screening and treatment was 2 weeks (±7 days).Efficacy and safety were evaluated at 4 weeks (±7 days), 8 weeks (±7 days) after treatment, and every 8 weeks (±7 days) thereafter.Once a subject develops disease progression (based on investigator evaluation or imaging evidence), the subject should discontinue the study.Cessation of treatment for any reason should be followed by a study end visit within 4 weeks (±7) days after the last study administration to collect information on all possible adverse events and drug combinations.Drug - related or possibly related adverse events should be followed up until they are stable or resolved.SAE should be documented within 30 days of study cessation.KN035 can be used for up to 2 years.

When desease progression is suspected, researchers are allowed to reconfirm disease progression after 4 weeks using irRECIST criteria.During the confirmation of disease progression, if the investigator decides that the subject should continue to receive KN035 treatment, the following criteria must be met:

The researchers assessed whether the subjects had benefited or were likely to continue to benefit:

①Subjects can tolerate study drug therapy;

②There were no medical events (e.g., central nervous system metastases) in which tumor progression was rapid or urgent intervention was required.

Study endpoint analysis will be performed when the last patient is followed for 24 weeks or disease progression or death is observed.If there is still no disease progression or intolerable adverse reactions, the patient will continue to receive KN035 treatment until the disease progression, death, occurrence of intolerable adverse reactions or treatment for 1 year (the researcher will give follow-up treatment recommendations according to the specific situation, if the original treatment is continued, the patient can still receive KN035 treatment for free).Treatment options after disease progression will be implemented at the discretion of the investigator.After the end of the study visit, subjects will enter the post-study follow-up period to collect survival data OS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 or above, 70 or below;
2. Patients with multiple primary tumors (currently suffering from colorectal cancer) diagnosed by histopathology (diagnostic criteria: ①the diagnosis of each malignant tumor must be confirmed by tissue/cytology;

   ②the pathological diagnosis of each malignant tumor has its unique pathological morphological support, different from other diagnoses;

   ③each malignant tumor diagnosis of the original site occurred in different parts, any two diagnosis is not mutually continuous;

   ④one of the diagnosis must be primary bowel cancer; (except for bowel cancer, other tumors do not need anti-tumor treatment);
3. Currently suffering from intestinal cancer and distant metastasis;
4. Received second-line or above treatment before, and the disease progress was determined by imaging; Or unable to tolerate any line treatment (including adjuvant or first-line treatment, etc., first-line treatment requires oxaliplatin, irinotecan and fluorouracil drugs);
5. At least one measurable lesion (RECIST 1.1);
6. ECOG score 0 or 1;
7. Expected survival≥12 weeks;
8. Adequate organ and bone marrow function (no hematopoietic growth factor, blood transfusion or platelet therapy was given within 1 week prior to the first study) :

(1) blood routine examination: leukocyte ≥3.0 ×109/L, neutrophil ≥1.5 ×109/L, platelet ≥75 ×109/L, hemoglobin ≥ 9.0g /dL; (2) liver function: total bilirubin ≤1.5 ×ULN; ALT/AST≤2.5 ×ULN without liver metastasis; ALT/AST≤5 ×ULN in liver metastasis; (3) renal function: serum creatinine≥1.5 x ULN; (4) adequate cardiac function, left ventricular ejection fraction (LVEF) > 50% of 2-d echocardiography.

9. Fully understand the study and sign informed consent voluntarily; 10. Women of reproductive age who have had a negative pregnancy test are willing to take effective contraceptive measures during the study period and within 90 days after the last dose of medication.

Exclusion Criteria:

1. Participate in clinical trials of other research drugs within 30 days before the first study drug treatment;Or received anti-tumor therapy within 2 weeks, including but not limited to chemotherapy, radiotherapy, targeted therapy, or anti-tumor therapy, the toxic response has not returned to the level 0 or level 1 (hair loss, ≤grade 2 peripheral neurotoxicity induced by chemotherapy can be included);
2. Previous immune checkpoint drug therapy;
3. Major surgery (except biopsy) or incomplete incision healing was performed within 4 weeks before the first study of drug therapy;
4. Ascites requiring drainage or diuretic treatment or hydrothorax or pericardial effusion requiring drainage and/or symptoms of shortness of breath within 2 weeks before the first study;
5. Active brain metastasis or spinal cord compression;For patients with brain metastasis who had received previous treatment, if the clinical conditions were stable within 4 weeks before the first study of drug treatment and the imaging evidence did not show the disease progression, and if they did not need corticosteroid treatment within 2 weeks before the first treatment, they could be considered to be enrolled.
6. Active, known or suspected autoimmune diseases (patients with vitiligo who do not require systematic treatment within 2 years before the first study of drug therapy are allowed to be enrolled;Patients with hypothyroidism requiring only thyroid hormone replacement therapy, type 1 diabetes requiring only insulin replacement therapy, and patients with pituitary inflammation and adrenocortical dysfunction requiring only physiological hormone replacement therapy can be enrolled);
7. Hiv-infected patients;
8. An active bacterial or fungal infection requiring systematic treatment 14 days before the first study drug treatment;
9. Previous history of interstitial lung disease, drug-induced interstitial lung disease, radioactive pneumonia, symptomatic interstitial lung disease, or any evidence of active pneumonia on chest CT scan within 4 weeks prior to initial study drug treatment;
10. HBV DNA≥2000 IU/ml (or 104 copies /ml) during screening period in patients with hepatitis b; Note: for enrolled subjects with anti-hbc (+)/HBsAg (+)/HBV DNA<2000 IU/ml or anti-hbc (+)/HBsAg (-)/HBV DNA<2000 IU/ml, antiviral therapy must be provided at the same time during the trial, either with the original drug or entecavir.For enrolled HCV rna-positive subjects, it was up to the investigator to decide whether to also receive antiviral therapy.
11. Clinically significant cardiovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina, cerebrovascular accident or transient ischemic attack, and congestive heart failure within the first 6 months of enrollment (New York heart association grade ≥ 2);Arrhythmias that require other antiarrhythmic drugs in addition to beta blockers or digoxin;Repeated electrocardiogram (ecg) detection of QTcF interval of >450 milliseconds (ms);Hypertension not well controlled by antihypertensive drugs (systolic blood pressure >150mmHg, diastolic blood pressure >100mmHg);
12. Abnormal thyroid function exists, and the use of drugs cannot maintain thyroid function in the normal range;
13. Clinically significant abnormal serum electrolyte level;
14. Immunosuppressive drugs were used within 2 weeks before the first study drug treatment, excluding local or systemic glucocorticoids not exceeding 10 mg/ d prednisone or other glucocorticoids of equivalent dose;
15. Live vaccine should be administered within 4 weeks before or during the first study period of drug therapy.
16. Has a history of severe allergic reactions to chimeric or human antibodies or fusion proteins or is known to be allergic to biological products or any component of KN035 produced from Chinese hamster ovary cells;
17. Pregnant or lactating women;
18. Fertility but unwillingness to accept effective contraception;
19. Any other disease, metabolic disorder or abnormal laboratory test, the researchers have reason to suspect that the patient is not fit to be treated with the study drug, or will affect the interpretation of the study results, or put the patient at high risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 1 year
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China